CLINICAL TRIAL: NCT03891940
Title: Evaluation of Changes of Swallowing Motor Function After Cervical Spine Surgery With Anterior Approach- the Implication of High Resolution Impedance Manometry
Brief Title: Swallowing Motor Function After Cervical Spine Surgery With Anterior Approach
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201901089RINC
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Patients Receiving Anterior Cervical Spine Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient receiving Anterior Cervical Spine Surgery: 1. Patients who fulfill the criteria of anterior cervical spine surgery under general anesthesia
  2. Aged from 20-80 years old
  Interventions: Procedure: patients recieving anterior cervical spine surgery

INTERVENTIONS:
Procedure: patients recieving anterior cervical spine surgery — Anterior cervical discectomy with fusion, or ACDF, is a surgery designed to relieve spinal cord or nerve root pressure in the neck by removing all or part of a damaged disc

SUMMARY:
Dysphagia is a well-known complication following anterior cervical spine surgery. However, which muscle at oropharyngeal region weakness and the recovery course of these patients are still unknown.

The ultrasonography was used to measure the oropharyngeal swallowing function. The high resolution impedance manometry (HRIM) could be used to measure the postoperative recovery esophageal function.

we aimed to observe the changes and recovery course swallowing function parameters during the preoperative and postoperative period in the patients receiving anterior cervical spine surgery by HRIM and ultrasonography.

DETAILED DESCRIPTION:
Dysphagia is a well-known complication following anterior cervical spine surgery. However, which muscle at oropharyngeal region weakness and the recovery course of these patients are still unknown.

The ultrasonography was used to measure the oropharyngeal swallowing function. The high resolution impedance manometry (HRIM) could be used to measure the postoperative recovery esophageal function.

We aimed to observe the changes and recovery course swallowing function parameters during the preoperative and postoperative period in the patients receiving anterior cervical spine surgery by HRIM and ultrasonography. Consecutive patients who will fulfill the criteria of cervical spine surgery patients under general anesthesia and aged >= 20 will be enrolled. The patients would receive the dysphagia questionnaire. All subjects would receive the swallowing function by ultrasonography and HRIM before the surgeries. The cough test was also measured. After the surgery, the patient would be followed the swallowing function in the postoperative one day, 1 week, and 1 months, 3 months (If needed) by HRIM and ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who fulfill the criteria of anterior cervical spine surgery under general anesthesia 2. Aged from 20-80 years old

Exclusion Criteria:

- 1. Major systemic disease, such as congestive heart failure, liver cirrhosis, end stage renal disease and malignancy.

2. Patients who have the risk of difficult ventilation or intubation. 3. pregnant women 4. coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fulfill the criteria of anterior cervical spine surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-26 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
upper esophageal sphincter pressure changes | everage 1 month in the perioperative period
  upper esophageal sphincter pressure changes measured by the HRIM

SECONDARY OUTCOMES:
hyoid bone movement | everage 1 month in the perioperative period
  the distance of hyoid bone movement measured by the ultrasonography

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai CJ, Cheng YJ, Lai DM, Wu CY, Chang WT, Tsuang FY. Applying High-Resolution Impedance Manometry for Detecting Swallowing Change in Anterior Cervical Spine Surgery Patients. Front Surg. 2022 Mar 16;9:851126. doi: 10.3389/fsurg.2022.851126. eCollection 2022. PMID 35372473